CLINICAL TRIAL: NCT04044716
Title: Nurse Initiated Auricular Acupressure for Post-operative Pain Management in Knee and Hip Arthroplasty Patients
Brief Title: Nurse Initiated Acupressure for Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00057513
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Results first posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Pain, Postoperative; Pain, Acute
Keywords: auricular acupressure; anesthesia
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Arm 1 Treatment group, Arm 2 Control group, Arm 3 Nurse Interventionist group
Who Masked: Outcomes Assessor
Masking Description: Statistician blinded to study arms during analysis phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Auricular acupressure Group (Experimental): The Auricular acupressure (AA) nurses will place the acupressure pellet pads on the participants in this group post-operatively.
  Interventions: Device: Auricular acupressure; Other: Standard of care pain management
- Standard of care Group (Active Comparator): Participants in this group will receive standard of care pain management by the treating physician.
  Interventions: Other: Standard of care pain management
- Nurse Interventionists (No Intervention): Nurses who were trained to apply the auricular acupressure pads/pellets in the the holding room prior to surgery.

INTERVENTIONS:
Device: Auricular acupressure — Trained nurses in auricular acupressure will place acupressure beads on 5 acupoints on each ear (cingulate gyrus, thalamus, omega-2, point zero, and Shen Men). The nurse will do the initial activation of the acupressure site by applying pressure for 30 seconds to each point until the participant reports tingling or moderate degree of pressure. Participant will be given instructions to do this three times a day for a total of 5 days. Acupoints were selected based on recommendation of faculty acupuncturist.
  Other Names: acupressure
  Arms: Auricular acupressure Group
Other: Standard of care pain management — The participant post-operative pain will be managed following the standard protocol by the treating physician.
  Arms: Auricular acupressure Group; Standard of care Group

SUMMARY:
The purpose of pilot study is to test the feasibility of nurse initiated post-operative bilateral auricular acupressure as an adjunct to medication for post-operative pain management.

DETAILED DESCRIPTION:
Postoperative pain management has become an area of concern over the last decade due to the opioid epidemic and concerns related to their use as the primary pain management strategy. Joint Commission requires that hospitals have additional pain non-pharmacologic pain management tools at their disposal to an effort decrease the reliance on opioids. Acupuncture and acupressure have been used for centuries in the management of a variety of disorders including pain. Unlike acupuncture, acupressure can be easily applied with limited training and is within the scope of practice for nurses, according to the North Carolina Board of Nursing. Thus evidence based non-pharmacologic strategies that can be deployed by nursing are of benefit to hospital organizations.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-80 admitted for knee or hip arthroplasty
* Pre-surgery morphine equivalent < 50
* American Society of Anaesthesiologists (ASA) score < 3

Exclusion Criteria:

* Participants with a history of skin disease (psoriasis), adhesive allergy, history of delirium, or cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn S Huffman, WHNP, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Davie Medical Center, Bermuda Run, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Auricular Acupressure Group: The Auricular acupressure (AA) nurses will place the acupressure pellet pads on the participant post-operatively.
  Auricular acupressure: Trained nurses in auricular acupressure will place acupressure beads on 5 acupoints on each ear (cingulate gyrus, thalamus, omega-2, point zero, and Shen Men). The nurse will do the initial activation of the acupressure site by applying pressure for 30 seconds to each point until the participant reports tingling or moderate degree of pressure. Participant will be given instructions to do this three times a day for a total of 5 days. Acupoints were selected based on recommendation of faculty acupuncturist.
  Standard of care pain management: The participant post-operative pain will be managed following the standard protocol by the treating physician.
Period: Overall Study
Arm/Group | Auricular Acupressure Group | Standard of Care Group | Nurse Interventionists
Started | 30 | 30 | 5
Completed | 27 | 27 | 5
Not Completed | 3 | 3 | 0
Not completed — participant stopped treatment but submitted partial data. | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: No baseline demographic information was gathered on participants in the Nurses arm, so those participants are not included in this section.
Groups:
- Total: Total of all reporting groups
Arm/Group | Auricular Acupressure Group | Standard of Care Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9.9) | 66 (8.3) | 66 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 27 | 29 | 56
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain). Pain score averaged across post-op days 1 - 4.
Time Frame: Up to Post-operatively day 4, at rising approximately 6 am
Population: 1 in Treatment and 2 in Standard of Care (SOC) group with incomplete missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 26 | 25
units on a scale | 3.03 (2.04) | 4.37 (2.18)
Statistical Analysis 1: Comparison: Auricular Acupressure Group vs Standard of Care Group; Test type: Superiority; p = .048, ANCOVA; age, joint involved in surgery, sex, baseline pain

2. Primary Outcome: Visual Analogue Pain Scale
Description: Average "pain before bed" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).Pain score averaged across post-op days 0 - 4.
Time Frame: Up to Post-operatively day 4, at the end of the day approximately 10 pm
Population: 3 in Treatment group and 3 in Standard of Care (SOC) group with missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 24 | 24
units on a scale | 5.27 (2.51) | 6.11 (2.21)
Statistical Analysis 1: Comparison: Auricular Acupressure Group vs Standard of Care Group; Test type: Superiority; p = 0.29, ANCOVA; adjusted for age, sex, type of surgery (joint), baseline pain

3. Primary Outcome: Medication Use - Outpatient Opioids
Description: Amount of medication use after discharge recorded in total morphine equivalent dose from discharge through day 4 postoperatively
Time Frame: Up to post-operatively day 4
Population: 1 in Treatment group and 1 in Standard of Care (SOC) group with missing data.
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 26 | 26
morphine milligram equivalents | 74.2 (58.9) | 88.6 (73.1)
Statistical Analysis 1: Comparison: Auricular Acupressure Group vs Standard of Care Group; Test type: Superiority; p = 0.64, ANCOVA; adjusted for age, sex, type of surgery (joint), baseline morphine milligram equivalents (MME)

4. Primary Outcome: Medication Use - Inpatient Opioids
Description: Amount of medication recorded in morphine equivalent dose while in hospital (not including anesthesia)
Time Frame: Up to post-operatively day 4
Population: Data obtained from hospital medication administration record on all participants.
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 30 | 30
MME | 37.8 (28.3) | 35.8 (28.6)
Statistical Analysis 1: Comparison: Auricular Acupressure Group vs Standard of Care Group; Test type: Superiority; p = 0.86, ANCOVA; adjusted for age, sex, type of surgery (joint), baseline MME, and time in hospital

5. Primary Outcome: Medication Use - Total Other Analgesics
Description: Amount of of other analgesics other than aspirin and not part of anesthesia record from immediate post-operative period to day 4 post-op in reported milligrams.
Time Frame: Up to post-operatively day 4
Population: 1 in Treatment group and 3 in Standard of Care (SOC) group with missing data.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 26 | 24
milligrams | 13643 (4615) | 13766 (3395)
Statistical Analysis 1: Comparison: Auricular Acupressure Group vs Standard of Care Group; Test type: Superiority; p = 0.661, ANCOVA — adjusted for age, type of surgery (joint), and sex

6. Secondary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 30 | 30
units on a scale | 2.30 (2.28) | 2.84 (2.69)

7. Secondary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).
Time Frame: post-operatively day 1, at rising
Population: Data from "other" participant in treatment group who stopped study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 28 | 27
units on a scale | 3.05 (2.36) | 3.90 (2.52)

8. Secondary Outcome: Visual Analogue Pain Scale
Description: Total score 0 to 10 on visual analogue scale, anchors 0=no pain, 10 equals worse pain.
Time Frame: post-operatively day 2, at rising
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 27 | 27
units on a scale | 3.76 (2.79) | 5.01 (2.70)

9. Secondary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).
Time Frame: post-operatively day 3, at rising
Population: 2 in Treatment with missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 25 | 27
units on a scale | 2.60 (2.02) | 4.46 (2.42)

10. Secondary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).
Time Frame: post-operatively day 4, at rising
Population: 2 in Treatment and 2 in Standard of Care (SOC) group with missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 25 | 25
units on a scale | 2.81 (2.13) | 4.25 (2.37)

11. Secondary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).
Time Frame: post-operatively day 1, at the end of the day
Population: 1 in Standard of Care group with missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 27 | 26
units on a scale | 5.64 (3.11) | 6.46 (2.54)

12. Secondary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).
Time Frame: post-operatively day 2, at the end of the day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 27 | 27
units on a scale | 5.79 (2.73) | 6.48 (2.41)

13. Secondary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).
Time Frame: post-operatively day 3, at the end of the day
Population: 2 in Treatment with missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 25 | 27
units on a scale | 4.78 (2.74) | 6.27 (2.49)

14. Secondary Outcome: Visual Analogue Pain Scale
Description: Average "pain upon awakening" score from 0 to 10 using visual analogue scale (0= no pain, 10= worst pain).
Time Frame: post-operatively day 4, at the end of the day
Population: 3 in Treatment and 3 in Standard of Care (SOC) group with missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 24 | 24
units on a scale | 4.47 (2.75) | 5.80 (2.46)

15. Secondary Outcome: Mean Number of Pellets Retained
Description: Mean number of pellets retained on post-operative day 4. This Outcome Measure was pre-specified to be assessed for the "Auricular Acupressure Group" Arm only.
Time Frame: Up to post-operatively day 4
Population: 3 in Treatment with missing data.
Measure: Mean (Standard Deviation); unit: number of pellets
Units Other Than Participants: Pellets
Arm/Group | Auricular Acupressure Group
Number analyzed (Participants) | 24
Number analyzed (Pellets) | 10
number of pellets | 7.38 (4.15)

16. Secondary Outcome: Number of Participants Who Responded They Were Satisfied With Pain Management
Description: Likert scale with a total score of 0 to 6--higher scores denotes worse outcomes. Force choice: very satisfied, satisfied, somewhat satisfied, somewhat dissatisfied, dissatisfied, very dissatisfied. Any degree of satisfaction compared to any degree of dissatisfaction. Satisfied included responses very satisfied to somewhat satisfied
Time Frame: post-operatively day 4
Population: 8 in Treatment and 5 in Standard of Care (SOC) group with missing data. Results indicate number of respondents who endorsed they were satisfied (very satisfied to somewhat satisfied) with pain management.
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 19 | 22
Participants | 19 | 21

17. Secondary Outcome: Number of Participants Who Responded "Yes, Would Definitely Consider Using in the Future."
Description: Participants were asked if they "would consider using auricular acupressure in the future for pain if recommended by a nurse or physician?" Possible answers are "no, would not use again", "maybe", or "Yes, would definitely consider using in the future."
Time Frame: post-operatively day 4
Population: 6 in Treatment and 5 in Standard of Care (SOC) group with missing data. Results are percent of total respondents who selected: "Yes, would definitely consider using in the future."
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupressure Group | Standard of Care Group
Number analyzed (Participants) | 21 | 22
Participants | 19 | 13

18. Secondary Outcome: Nurse Time to Deploy Pellets
Description: Reported as the number of minutes that it took nurse interventionists to place acupressure seeds (pellets), activate, and provide instruction.
Time Frame: post-operatively day 5
Population: Data collected while inpatient on all 30 participants in treatment arm. Missing data on 2 participants. This outcome applies to the AA group only.
Measure: Median (Full Range); unit: minutes
Arm/Group | Auricular Acupressure Group
Number analyzed (Participants) | 28
minutes | 13.5 [6 to 18]

19. Secondary Outcome: Number of Nurse Concerns Reported
Description: Review nurse reports in encounters. Count number of concerns pooled across all participants in encounters with disruption of workflow due to care unit or patient barriers documented while participant was in hospital. Concerns included workflow and patient barriers. This outcome applies to nurse interventionists arm only.
Time Frame: post-operatively day 0 and 1
Measure: Number; unit: number of concerns reported
Units Other Than Participants: encounters
Arm/Group | Nurse Interventionists
Number analyzed (Participants) | 5
Number analyzed (encounters) | 120
number of concerns reported | 10

ADVERSE EVENTS:
Time Frame: Adverse events collected from post-operative day 0 - post-operative day 5
Description: self reported on daily study questionnaire; no adverse event information gathered for Nurse Interventionist arm
Arm/Group | Auricular Acupressure Group | Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auricular Acupressure Group (N=30) | Standard of Care Group (N=30)
Irritation at auricular acupressure site (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT04044716/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04044716/ICF_000.pdf